CLINICAL TRIAL: NCT02909907
Title: Comparison of Botulinum Toxin Injections in Forearm FLexor Plus EXtensor Muscles Versus Flexor Muscles Alone for the Treatment of Essential Hand Tremor (FLEX-D ET)
Brief Title: Comparison of Botulinum Toxin Injections in Forearm FLexor Plus EXtensor Muscles vs. Flexor Muscles Alone for Treatment of Essential Hand Tremor(FLEX-D ET)
Acronym: FLEX-D ET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-1519
Record Dates: First submitted 2016-08-11; First posted 2016-09-21 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor | interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 150 units of abobotulinumtoxinA (Experimental): 150 units of abobotulinumtoxinA in flexor compartment of dominant arm (75 units in flexor carpi radialis [FCR] and 75 units in flexor carpi ulnaris [FCU]) along with placebo in extensor carpi radialis (ECR) and extensor carpi ulnaris (ECU)
  Interventions: Drug: Botulinum toxin; Other: Placebo
- 75 units of abobotulinumtoxinA (Experimental): 75 units of abobotulinumtoxinA in FCR and FCU and 25 units in ECR and ECU
  Interventions: Drug: Botulinum toxin

INTERVENTIONS:
Drug: Botulinum toxin — Botulinum injections into dominant upper extremity using protocol outlined above.
  Other Names: BoNT
Other: Placebo — Placebo injections in extensor carpi radialis (ECR) and extensor carpi ulnaris (ECU) per protocol outlined above
  Arms: 150 units of abobotulinumtoxinA

SUMMARY:
To compare the efficacy of botulinum toxin (BoNT) injections in forearm flexors plus extensor muscles versus flexors alone for the treatment of essential hand tremor (ET).

DETAILED DESCRIPTION:
The investigators propose a pilot, single center, double blind, randomized, parallel, placebo controlled trial comparing 2 (BoNT) injection patterns for treatment of moderate to severe essential tremor. The investigators will recruit 20 patients with (ET).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and over, male or female patient with (ET) involving at least their dominant hand, as diagnosed by a movement disorders neurologist.
2. Having bothersome hand tremor in dominant hand with a hand TRS ≥2
3. On stable medications during last 30 days prior to enrollment.

Exclusion Criteria:

1. Presence of secondary causes of tremor, such as dystonia and parkinsonism
2. Any contraindication to botulinum toxin injections (e.g. motor neuron disease, neuromuscular junction disease, etc.)
3. History of surgical treatment for (ET).
4. Dementia as defined by DSM-V criteria
5. Patients with suboptimally treated depression and significant depressive symptoms as defined by a PHQ-9 score of ≥15 (PHQ-9 scores 1-4 Minimal depression; 5-9 Mild depression; 10-14 Moderate depression; 15-19 Moderately severe depression; 20-27 Severe depression). Antidepressant medications, prescribed for depression or anxiety, will be allowed if the patient has been on a stable dose for at least 30 days.
6. Patients with suboptimally treated anxiety and significant anxiety symptoms as defined by a GAD-7 score of ≥15 (GAD-7 scores 0-4: minimal anxiety; 5-9: mild anxiety; 10-14: moderate anxiety; 15-21: severe anxiety). Anti-anxiety medications, prescribed for anxiety, will be allowed if the patient has been on a stable dose for at least 30 days.
7. Significant renal, hepatic, cardiac and thyroid disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-08; Primary Completion 2018-02 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Fernandez, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 12-week, pilot, randomized (1:1 ratio), double-blind, placebo-controlled study of 21 patients with ET evaluated by a movement disorders specialist at the Cleveland Clinic.
Pre-assignment Details: Twenty-one patients were enrolled to participate, but one patient was removed from the sample due to being an extreme outlier on most outcomes of interest, and another patient dropped out after the baseline visit.
Groups:
- Flexors Alone: 75 units of abobotulinumtoxinA in FCR and FCU and 25 units in ECR and ECU
  Botulinum toxin: Botulinum injections into dominant upper extremity using protocol outlined above.
- Flexors Plus Extensors: 150 units of abobotulinumtoxinA in flexor compartment of dominant arm (75 units in flexor carpi radialis [FCR] and 75 units in flexor carpi ulnaris [FCU]) along with placebo in extensor carpi radialis (ECR) and extensor carpi ulnaris (ECU)
  Botulinum toxin: Botulinum injections into dominant upper extremity using protocol outlined above.
  Placebo: Placebo injections in extensor carpi radialis (ECR) and extensor carpi ulnaris (ECU) per protocol outlined above
Period: Overall Study
Arm/Group | Flexors Alone | Flexors Plus Extensors
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flexors Alone | Flexors Plus Extensors | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (12.0) | 64.9 (9.1) | 69.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Right-handed [Number; unit: participants] | 9 | 7 | 16
TRS mean [Mean (Standard Deviation); unit: units on a scale] — TRS: Tremor Rating Scale : scale composed of 6 items rated from 0-4. 0=none or normal and 4 = very severe or high level of disability. Total score is the sum of all items. Max score 24 ( maximal severity of tremor) Minimal score 0= no tremor/normal.
  units on a scale | 12.9 (4.6) | 11.3 (4.1) | 12.1 (4.3)
QUEST Health status self-report, med(IQR) [Mean (Inter-Quartile Range); unit: units on a scale] — QUEST ( Quality of life in Essential tremor Questionnaire )
  Heath Status:
  In general, how would you rate your overall health? (0=very poor health, 100=excellent/perfect health)
  Circle: 0 5 10 15 20 25 30 35 40 45 50 55 60 65 70 75 80 85 90 95 100
  units on a scale | 82.5 [75 to 90] | 82.5 [75 to 90] | 82.5 [75 to 90]
QUEST Quality of Life self-report, mean(SD) [Mean (Standard Deviation); unit: units on a scale] — Quality of Life in Essential Tremor Questionnaire (QUEST)
  Overall Quality of Life:
  Overall, how would you rate your quality of life? (0=very poor health, 100=excellent/perfect health):
  Circle: 0 5 10 15 20 25 30 35 40 45 50 55 60 65 70 75 80 85 90 95 100
  units on a scale | 84 (9.7) | 82.8 (6.7) | 83.4 (8.2)
QUEST Communication, med (IQR) [Median (Inter-Quartile Range); unit: units on a scale] — Quality of Life in Essential Tremor Questionnaire (QUEST): Dimension Communication: total questions 3 Possible answers: Each answer correspond to a numeric value : N=0 R=1 S=2 F=3 A=4 NA=blank N = Never/Not applicable R = Rarely S = Sometimes F = Frequently A = Always/Yes Scoring Algorithm: Total applicable points for each dimension/total possible points ( # of applicable questionsx 4 ) for each dimension X100 = dimension score.
  Maximal Score 100=worse quality of life due to tremor. Minimal score 0= Best quality of life.
  units on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
QUEST Work, med (IQR) [Median (Inter-Quartile Range); unit: units on a scale] — Quality of Life in Essential Tremor Questionnaire (QUEST): Dimension Work: total questions 6 Possible answers: Each answer correspond to a numeric value : N=0 R=1 S=2 F=3 A=4 NA=blank N = Never/Not applicable R = Rarely S = Sometimes F = Frequently A = Always/Yes Scoring Algorithm: Total applicable points for each dimension/total possible points ( # of applicable questionsx 4 ) for each dimension X100 = dimension score.
  Maximal Score 100=worse quality of life due to tremor. Minimal score 0= Best quality of life.
  units on a scale | 0 [0 to 8.3] | 8.3 [0 to 25] | 0 [0 to 12.5]
QUEST Hobbies, med (IQR) [Median (Inter-Quartile Range); unit: units on a scale] — Quality of Life in Essential Tremor Questionnaire (QUEST): Dimension Hobbies: total questions 3 Possible answers: Each answer correspond to a numeric value : N=0 R=1 S=2 F=3 A=4 NA=blank N = Never/Not applicable R = Rarely S = Sometimes F = Frequently A = Always/Yes Scoring Algorithm: Total applicable points for each dimension/total possible points ( # of applicable questionsx 4 ) for each dimension X100 = dimension score.
  Maximal Score 100=worse quality of life due to tremor. Minimal score 0= Best quality of life.
  units on a scale | 0 [0 to 8.3] | 0 [0 to 50] | 0 [0 to 50]
QUEST Physical, med (IQR) [Median (Inter-Quartile Range); unit: units on a scale] — Quality of Life in Essential Tremor Questionnaire (QUEST): Dimension Physical: total questions 9 Possible answers: Each answer correspond to a numeric value : N=0 R=1 S=2 F=3 A=4 NA=blank N = Never/Not applicable R = Rarely S = Sometimes F = Frequently A = Always/Yes Scoring Algorithm: Total applicable points for each dimension/total possible points ( # of applicable questionsx 4 ) for each dimension X100 = dimension score.
  Maximal Score 100=worse quality of life due to tremor. Minimal score 0= Best quality of life.
  units on a scale | 44.4 [33.3 to 72.2] | 61.1 [58.3 to 61.1] | 61.1 [33.3 to 72.2]
QUEST Psychosocial, med (IQR) [Median (Inter-Quartile Range); unit: units on a scale] — Quality of Life in Essential Tremor Questionnaire (QUEST): Dimension Communication: total questions 9 Possible answers: Each answer correspond to a numeric value : N=0 R=1 S=2 F=3 A=4 NA=blank N = Never/Not applicable R = Rarely S = Sometimes F = Frequently A = Always/Yes Scoring Algorithm: Total applicable points for each dimension/total possible points ( # of applicable questionsx 4 ) for each dimension X100 = dimension score.
  Maximal Score 100=worse quality of life due to tremor. Minimal score 0= Best quality of life.
  units on a scale | 8.3 [0 to 25] | 25 [11 to 41.7] | 11.1 [8.3 to 30.5]
QUEST Summary Index, med (IQR) [Mean (Inter-Quartile Range); unit: units on a scale] — Quality of Life in Essential Tremor Questionnaire: Total summary index
  30-item, ET-specific quality of life scale
  Items contribute to 5 dimensions: Physical/ADL, Psychosocial, Communication, Hobbies/Leisure, and Work/Finances. The score on each scale is a percentage of the total score possible, a higher score indicates greater dissatisfaction with that domain.
  The total summary index corresponds to the mean of the five domain scores. Maximal score 100: worse quality of life. Minimal Score 0: best quality of life.
  units on a scale | 12.2 [10.6 to 20] | 26.4 [17.8 to 29.4] | 17.8 [11.1 to 29.4]
PHQ-9, med (IQR) [Median (Inter-Quartile Range); unit: units on a scale] — Patient Health Questionnaire - 9 PHQ-9
  9 question items scored from : 0=not at all , 1= Several Days, 2=More than half the days, 3=nearly every day .
  Total score is the sum of all items.
  Interpretation of Total Score Total Score Depression Severity 0-4 Minimal depression 5-9 Mild depression 10-14 Moderate depression 15-19 Moderately severe depression 20-27 Severe depression
  Minimum score: 0 : no depression. Maximal Score 27 : severe depression.
  units on a scale | 0.5 [0 to 6] | 4 [1 to 7] | 2 [0 to 6]
GAD-7, med (IQR) [Median (Inter-Quartile Range); unit: Score on a scale] — Generalized Anxiety Disorder 7 item ( GAD-7)
  Total of 7 questions scored from 0=not at all , 1= several days, 2= More than half the days, 3= Nearly every day.
  Total score = total sum of all items. Maximal score=21, minimal Score =0
  Interpretation of the score:
  > or = 10 probable diagnosis of Generalized anxiety disorder, Confirm by further evaluation.
  0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety
  Score on a scale | 0 [0 to 1] | 2 [0 to 3] | 0 [0 to 3]
Age of onset, med (IQR) [Median (Inter-Quartile Range); unit: years] | 55.5 [25 to 73] | 58 [40 to 64] | 58 [30 to 68]
Disease duration, med (IQR) [Median (Inter-Quartile Range); unit: Years] | 5.5 [2 to 42] | 5 [2 to 10] | 5 [2 to 16]
Main Grip Strength [Median (Inter-Quartile Range); unit: Kg] | 30.8 [22.7 to 36.7] | 28 [26.7 to 33.3] | 29.7 [23.7 to 36.7]

OUTCOME MEASURES:

1. Primary Outcome: Difference in the 6 Week Post Injection Patient Global Impression of Improvement Scale (PGIS) Between Flexors Along and Flexors Plus Extensors Groups.
Description: 6 weeks post injection Clinician Global Impression if improvement Scale (CGIS)
  Assessment of improvement graded by the patient on a -4 to +4 scale
  * -4 = severe worsening
  * 0 = no change
  * +4 = complete abolishment of symptoms
  Higher scores represent better outcome.
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Flexors Alone | Flexors Plus Extensors
Number analyzed (Participants) | 10 | 9
score on a scale | 1.2 [1 to 3] | 2.2 [1.6 to 4]

2. Secondary Outcome: Difference in Tremor Rating Scale Score (TSR)Change From Baseline to Week 6 Between Flexors Alone and Flexors Plus Extensors Groups.
Description: TRS: Tremor Rating Scale : scale composed of 6 items rated from 0-4. 0=none/normal and 4 = very severe/high level of disability. Total score is the sum of all items. Max score 24 ( maximal severity of tremor) Minimal score 0= no tremor/normal.
Time Frame: Baseline and 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Flexors Alone | Flexors Plus Extensors
Number analyzed (Participants) | 10 | 9
score on a scale | -5 [-6 to -4] | -5 [-6 to -4]

3. Secondary Outcome: Difference in the 6 Week Post Injection Clinician Global Impression of Improvement Scale (CGIS) Between Flexors Along and Flexors Plus Extensors Groups.
Description: 6 weeks post injection Clinician Global Impression if improvement Scale (CGIS)
  Assessment of improvement graded by clinician on a -4 to +4 scale
  * -4 = severe worsening
  * 0 = no change
  * +4 = complete abolishment of symptoms
  Higher scores represent better outcome.
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Flexors Alone | Flexors Plus Extensors
Number analyzed (Participants) | 10 | 9
score on a scale | 1 [0 to 2] | 3 [1 to 3]

4. Secondary Outcome: Difference of the Quality of Life in Essential Tremor Questionnaire (QUEST) Summary Index Change at Week 6 Compared to Baseline Between Wrist Flexors Versus Wrist Flexors Plus Extensors Group.
Description: QUEST( Quality of Life in Essential Tremor Questionnaire ) is a 30-item, ET-specific quality of life scale . Items contribute to five dimensions. Physical/ADL (9 items ), Psychosocial (9 items), Communication (3 items), Hobbies/Leisure (3 items), and Work/Finances (6 items). The score on each scale is expressed as a percentage of the total score possible, with a higher score indicating greater dissatisfaction with that domain of QOL. A total or summary index corresponds to the mean of the five domain scores. The total summary index corresponds to the mean of the five domain scores. Maximal score 100: worse quality of life. Minimal Score 0: best quality of life. This outcome represents the median of the differences between baseline and week 6 in QUEST summary index.Positive index change values indicate that the score increased and negative values indicate that the score decreased.
Time Frame: Baseline and 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Flexors Alone | Flexors Plus Extensors
Number analyzed (Participants) | 10 | 9
score on a scale | 1.1 [-1.7 to 5.6] | -5.3 [-6.11 to 1.1]

5. Secondary Outcome: Difference in the Post Injection Grip Strength Change Between Flexor Only Group and Flexor and Extensors Group at 6 Weeks.
Description: the median of the differences in grip strength between baseline and week 6, A negative value indicates a decrease in grip strength in Kg at week 6.
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: Kilograms
Arm/Group | Flexors Alone | Flexors Plus Extensors
Number analyzed (Participants) | 10 | 9
Kilograms | -6.2 [-15.3 to -5.3] | -11 [-13.3 to 7.3]

6. Secondary Outcome: 12 Weeks Post Injection Tremor Rating Scale for Flexors Group and Flexors Plus Extensors Group.
Description: TRS: Tremor Rating Scale : scale composed of 6 items rated from 0-4. 0=none or normal and 4 = very severe or high level of disability. Total score is the sum of all items. Max score 24 ( maximal severity of tremor) Minimal score 0= no tremor/normal.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Flexors Alone | Flexors Plus Extensors
Number analyzed (Participants) | 10 | 9
score on a scale | 6 [6 to 9] | 6 [3 to 12]

7. Secondary Outcome: 12 Week Post Injection in Clinician Global Impression Scale-Improvement Subscale (CGIS)
Description: 12 week post injection in Clinician Global Impression Scale-Improvement Subscale (CGIS)
  Assessment of improvement graded by the clinician on a -4 to +4 scale
  * -4 = severe worsening
  * 0 = no change
  * +4 = complete abolishment of symptoms
  Higher scores represent better outcome.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Flexors Alone | Flexors Plus Extensors
Number analyzed (Participants) | 10 | 9
score on a scale | 3 [1 to 3] | 3 [1 to 3]

8. Secondary Outcome: 12 Week Post Injection Patient Global Impression Scale-Improvement Subscale (PGIS)
Description: Patient Global Impression Scale-Improvement Subscale (PGIS)
  Assessment of improvement graded by patient on a -4 to +4 scale
  * -4 = severe worsening
  * 0 = no change
  * +4 = complete abolishment of symptoms
  Higher scores represent better outcome.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Flexors Alone | Flexors Plus Extensors
Number analyzed (Participants) | 10 | 9
score on a scale | 1 [1 to 3] | 3 [1 to 3]

9. Secondary Outcome: Difference of Quality of Life in Essential Tremor Questionnaire (QUEST) Summary Index Change at Week 12 Compared to Baseline Between Wrist Flexors Versus Wrist Flexors Plus Extensors Group.
Description: QUEST( Quality of Life in Essential Tremor Questionnaire ) is a 30-item, ET-specific quality of life scale . Items contribute to five dimensions. Physical/ADL (9 items ), Psychosocial (9 items), Communication (3 items), Hobbies/Leisure (3 items), and Work/Finances (6 items). The score on each scale is expressed as a percentage of the total score possible, with a higher score indicating greater dissatisfaction with that domain of QOL. A total or summary index corresponds to the mean of the five domain scores. The total summary index corresponds to the mean of the five domain scores. Maximal score 100: worse quality of life. Minimal Score 0: best quality of life. This outcome represents the median of the differences between baseline and week 6 in QUEST summary index. Positive index change values indicate that the score increased and negative values indicate that the score decreased.
Time Frame: Baseline and 12 weeks.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Flexors Alone | Flexors Plus Extensors
Number analyzed (Participants) | 10 | 9
score on a scale | -1.67 [-3.9 to -0.56] | 0 [-6.11 to 6.67]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Flexors Alone | Flexors Plus Extensors
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 4/10 | 5/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flexors Alone (N=10) | Flexors Plus Extensors (N=9)
Finger Weakness (Nervous system disorders) | 4 | 5 — Weakness of fingers

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-02): https://cdn.clinicaltrials.gov/large-docs/07/NCT02909907/Prot_SAP_000.pdf